CLINICAL TRIAL: NCT00911872
Title: EVOLENCE® Assessment of Recovery Time and Impact of Dermal Filler Selection: The E-ART™ Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solish, Nowell, M.D. (Individual)
Responsible Party: Dr. Nowell Solish, Private Practice
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-ART
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2009-06-02 (Estimated); Status verified 2009-05

CONDITIONS: Aging
Keywords: wrinkles; dermal filler; collagen; soft tissue augmentation; aesthetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aging (Experimental)
  Interventions: Device: collagen (EVOLENCE)

INTERVENTIONS:
Device: collagen (EVOLENCE) — injectable collagen
  Other Names: EVOLENCE and EVOLENCE BREEZE

SUMMARY:
The purpose of this study is to gather information about the immediate effects and recovery time for treatment with EVOLENCE/EVOLENCE BREEZE for soft tissue augmentation. The time it takes for patients to feel comfortable with the results, and return to their normal daily routine is also of important interest

DETAILED DESCRIPTION:
The primary objective of this Investigator Initiated Study is to document recovery time/return to daily activities following facial soft-tissue augmentation with an EVOLENCE dermal filler. In addition, the immediate effects such as swelling, bleeding, bruising will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female > 18 years of age
* Need for soft tissue augmentation as evidenced by any of the following:

  * Bilateral-aging defects > 1 on the Modified Fitzpatrick Wrinkle Scale
  * Decrease in soft tissue volume in other areas of the face

Exclusion Criteria:

* History of positive hypersensitivity to porcine collagen-based products History of multiple food, drug, and substance allergies Autoimmune or collagen vascular disease Facial tissue augmentation within 6 months (HA) or 12 months Evolence/Evolence Breeze Botulinum-toxin A within 6 weeks Ablative laser treatments within 12 months Permanent facial implants Investigational product use within 30 days Pregnant and/or nursing woman or woman who plan to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Is to document recovery time/return to daily activities following facial soft-tissue augmentation with an EVOLENCE dermal filler | 7 Days

SECONDARY OUTCOMES:
the immediate effects such as swelling, bleeding, bruising will be assessed | 7 Days

CONTACTS AND LOCATIONS:
Overall Officials: Nowell Solish, MD, Principal Investigator — Private Practice
Locations (1):
- Nowell Solish Private Practice, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Solish NJ. Assessment of recovery time for the collagen products Dermicol-P35 27G and 30G. J Am Acad Dermatol. 2010 May;62(5):824-30. doi: 10.1016/j.jaad.2009.08.016. PMID 20398812